CLINICAL TRIAL: NCT03933631
Title: A Prospective Randomized Control Trial of Pilocarpine Use After Combined Cataract/Kahook Dual Blade Surgery
Brief Title: Pilocarpine Use After Kahook Goniotomy
Acronym: PAACK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-9829
Record Dates: First submitted 2019-04-26; First posted 2019-05-01 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma
Keywords: Cataract; Glaucoma Surgery; Vision; Cataract Surgery; Eye surgery
MeSH Terms: conditions — Glaucoma; Cataract | interventions — Pilocarpine; Prednisolone; prednisolone acetate; Ofloxacin

STUDY DESIGN:
Intervention Model Description: The "Treatment Group" will use 2% pilocarpine in the postoperative period in addition to standard postoperative drops (Prednisolone acetate and Ofloxacin). The "Control Group" will use only Prednisolone acetate and Ofloxacin, without pilocarpine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pilocarpine, Prednisolone acetate and Ofloxacin (Experimental): This group will use 2% pilocarpine in the postoperative period, for one month, in addition to standard postoperative drops (Prednisolone acetate and Ofloxacin)
  Interventions: Drug: Pilocarpine; Drug: Prednisolone; Drug: Ofloxacin
- Prednisolone acetate and Ofloxacin (standard of care) (Active Comparator): This group will use only the standard Prednisolone acetate and Ofloxacin, without pilocarpine.
  Interventions: Drug: Prednisolone; Drug: Ofloxacin

INTERVENTIONS:
Drug: Pilocarpine — pilocarpine hydrochloride ophthalmic solution 2% (20 mg/mL)
  Other Names: Isopto®
  Arms: Pilocarpine, Prednisolone acetate and Ofloxacin
Drug: Prednisolone — Prednisolone acetate ophthalmic suspension 1%
  Other Names: Pred Forte
Drug: Ofloxacin — Ofloxacin Drops
  Other Names: Ocuflox; Floxin

SUMMARY:
The goal of this study is to determine whether using pilocarpine provides added benefit to the success of combined cataract + Kahook Dual Blade (KDB) surgery.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness worldwide, and its treatment consists of lowering intraocular pressure to prevent damage to the optic nerve and loss of vision. Current methods for lowering intraocular pressure (IOP) include topical and oral medications, laser trabeculoplasty, microincisional glaucoma surgery (MIGS), and traditional incisional surgeries such as trabeculectomy and aqueous tube shunts. MIGS have become more popular in recent years as less invasive methods than traditional surgeries that effectively reduce IOP and help reduce the medication burden on patients. There are multiple available MIGS procedures, most of which act by increasing trabecular outflow. One such procedure is the goniotomy via Kahook Dual Blade (KDB), which is usually performed in combination with cataract surgery. KDB is an FDA approved device used to perform a goniotomy via an internal approach. Strips of the nasal angle trabecular meshwork are removed providing a direct pathway for aqueous outflow from the anterior chamber into the collector channels.

Pilocarpine, a parasympathomimetic agent, is a glaucoma medication that works by causing contraction of the ciliary muscle leading to opening of the trabecular meshwork. Due to its frequent dosing requirement and large number of ocular and systemic side effects, pilocarpine has largely fallen out of favor for the treatment of primary open angle glaucoma (POAG), except in patients for whom few other alternatives exist. However, pilocarpine is often used after goniotomy surgery. The rationale for its use after goniotomy procedure is for its miotic effect, which theoretically may prevent the formation of peripheral anterior synechiae. Formation of peripheral anterior synechiae can lead to the closure of the cleft that is generated and the possibility of failure of the procedure. While the theoretical benefit of pilocarpine has been proposed, its actual benefit has never been proven. This study will evaluate whether goniotomy via KDB / Cataract surgery without pilocarpine is non-inferior to the same surgery procedure followed by treatment with pilocarpine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ocular hypertension or open angle glaucoma undergoing combined cataract surgery with KDB in a single surgical center at Montefiore Medical Center with a single provider

Exclusion Criteria:

* Patients with previous history of eye surgeries (including laser procedures)

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with lowering of intraocular pressure (IOP) | From baseline to 1 year following procedure
  The percentage of patients who had a reduction in IOP of 20% or more from baseline will be summarized by study arm using descriptive statistics.

SECONDARY OUTCOMES:
Proportion of patients whose regimen was reduced by 1 medication or more | Up to 1 year following procedure
  The proportion/percentage of patients whose regimen was reduced by 1 medication or more during each routine post-operative monitoring visit following the combined cataract and KDB surgery procedure will be summarized by study arm using descriptive statistics.
Hypotensive medications | Up to 1 year following procedure
  The number and type of ocular hypotensive medications used following the procedure will be summarized by study arm using descriptive statistics.
Rate of progression towards further glaucoma surgery - Humphrey Visual Fields (HVF) | Up to 1 year following procedure
  The rate of progression towards additional glaucoma surgeries will be assessed using Humphrey Visual Fields (HVF) testing. Automated HVF testing will be used to detect and monitor the progression of glaucoma by mapping the patient's peripheral vision and detecting areas of vision loss. The rate of progression is assessed through software that assesses both trend and event analysis. Software trend analysis will be used to quantify how much vision is lost up to 1 year. Visual field loss rate will be summarized by study arm and reported using descriptive statistics.
Rate of progression towards further glaucoma surgery - Optical Coherence Tomography (OCT) | Up to 1 year following procedure
  The rate of progression towards additional glaucoma surgery will also be assessed using OCT scanning. OCT scanning will be used to obtain a quantitative measurement of structural of the retinal nerve fiber layer over time. OCT can reveal structural changes that often precede functional visual field loss and be an earlier indicator of progression. The rate of structural loss over time as measured by change in retinal nerve fiber thickness will be summarized and reported by study arm and reported using descriptive statistics.
Need for additional glaucoma surgery | Up to 1 year following procedure
  The need for additional glaucoma surgery will be determined by the number of patients who require additional glaucoma surgery following the scheduled cataract and KDB surgery. The number/percentage of patients requiring additional glaucoma surgery will be summarized by study arm using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jeng (Melissa) Yao, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Montefiore Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu K, Gazzard G, Bunce C, Wormald R. Ab interno trabecular bypass surgery with Trabectome for open angle glaucoma. Cochrane Database Syst Rev. 2016 Aug 15;(8):CD011693. doi: 10.1002/14651858.CD011693.pub2. PMID 27526051
- [Background] Johnson M. 'What controls aqueous humour outflow resistance?'. Exp Eye Res. 2006 Apr;82(4):545-57. doi: 10.1016/j.exer.2005.10.011. Epub 2006 Jan 4. PMID 16386733
- [Background] Seibold LK, Soohoo JR, Ammar DA, Kahook MY. Preclinical investigation of ab interno trabeculectomy using a novel dual-blade device. Am J Ophthalmol. 2013 Mar;155(3):524-529.e2. doi: 10.1016/j.ajo.2012.09.023. Epub 2012 Dec 4. PMID 23218696
- [Background] Swaminathan SS, Monsalve P, Zhou XY, Enriquez-Algeciras M, Bhattacharya SK, Dubovy SR, Junk AK. Histologic Analysis of Trabecular Meshwork Obtained From Kahook Dual Blade Goniotomy. Am J Ophthalmol. 2018 Aug;192:198-205. doi: 10.1016/j.ajo.2018.05.028. Epub 2018 Jun 5. PMID 29883587